CLINICAL TRIAL: NCT05231200
Title: Alberta (AB) Collaborative Quality Improvement Strategies to Improve Outcomes of Preterm Infants 32 - 36 Weeks' Gestation: A Stepped-Wedge Cluster Randomized Trial
Brief Title: Alberta Collaborative QI Strategies to Improve Outcomes of Moderate and Late Preterm Infants (ABC-QI Trial)
Acronym: ABC-QI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other); Alberta Health services (Other); Covenant Health, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-1336; 462647 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2022-01-06; First posted 2022-02-09 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Length of Stay
Keywords: Preterm infants; Evidence-based Practice for Improving Quality; Neonatal intensive care units

STUDY DESIGN:
Intervention Model Description: A stepped-wedge cluster randomized trial (SW-CRT) design. Each of the 12 participating NICUs (10 Level II and 2 Level III) are considered clusters and will be randomized to transition to the intervention arm at one of three-time points over a period of four years. The first year will be a baseline period where no clusters are exposed to the intervention. Based on the randomization, four NICUs will transition to the intervention arm at the end of each year. All clusters will have transitioned to the intervention arm by the start of year four.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm- Current management (Active Comparator): NICUs in the control arm can continue conducting QI activities relevant to current practice and current standard of care, but without receiving the interventions until they transition to the intervention arm.
  Interventions: Other: Current practice- standard of care
- Intervention Arm- Collaborative Quality implementation Strategies (Experimental): The study intervention is a constellation of collaborative QI strategies: 1) QI Team Building; 2) QI Education; 3) Implementation of 2 standardized practice care bundles (Respiratory Care, and Nutritional Care); 4) QI mentoring; and 5) Collaborative networking.
  Interventions: Behavioral: QI Team Building; Behavioral: QI education; Other: Standardized care bundle- respiratory care; Other: Standardized care bundle- nutritional care; Behavioral: QI mentoring; Behavioral: Collaborative networking

INTERVENTIONS:
Behavioral: QI Team Building — Each NICU will create a core QI team composed of 6-8 multidisciplinary members including a parent advisor, when feasible. This team will lead the QI activities and education, and champion the culture and practice change in the unit.
  Arms: Intervention Arm- Collaborative Quality implementation Strategies
Behavioral: QI education — Each NICU QI team will receive standardized QI education using the 6-hour EPIQ Workshop which involves hands-on approach to enable teams to successfully implement QI projects together. EPIQ 10 Steps and QI Tools will be used to build the team's understanding of QI using realistic improvement opportunities based on the standardized care bundles identified in the trial.
  Arms: Intervention Arm- Collaborative Quality implementation Strategies
Other: Standardized care bundle- respiratory care — A care bundle is a small, simple set (3-5 elements) of evidence-based practices that, when performed collectively and reliably, will result in improved patient outcomes. This bundle will aim to implement best practices for stabilization and respiratory care in moderate and late preterm infants (MLPIs) including
  1. establishing effective ventilation in the delivery room
  2. prevention of hypothermia
  3. early diagnosis and management of respiratory distress with continuous positive airway pressure (CPAP)
  4. standardized approach for surfactant indications and administration
  5. standardized approach for early extubation.
  Arms: Intervention Arm- Collaborative Quality implementation Strategies
Other: Standardized care bundle- nutritional care — A care bundle is a small, simple set (3-5 elements) of evidence-based practices that, when performed collectively and reliably, will result in improved patient outcomes. This bundle will aim to implement best practices for nutritional support in MLPIs including
  1. early initiation of enteral or parenteral nutrition;
  2. standardized tables for feeding initiation and progression
  3. optimizing breastfeeding and use of mother's own milk
  4. standardized approach for a transition from enteral nutrition via tube feeds to oral feeds.
  Arms: Intervention Arm- Collaborative Quality implementation Strategies
Behavioral: QI mentoring — Each NICU in the intervention arm will have one or more assigned members of the study team who are experienced in collaborative QI and EPIQ methods. The mentors will help local QI teams to engage frontline staff in QI and navigate the unit-specific challenges.
  Arms: Intervention Arm- Collaborative Quality implementation Strategies
Behavioral: Collaborative networking — The study team will conduct virtual meetings every 2 months for the NICUs in intervention arm allowing local QI teams to discuss progress, and share data. The investigators will arrange annual in-person or virtual meetings for the NICUs in the intervention arm to present projects, successes, and lessons learned. These NICUs will have continuing access to the data and will receive quarterly reports using statistical process control charts outlining the unit's performance compared to other units and to the group average.
  Arms: Intervention Arm- Collaborative Quality implementation Strategies
Other: Current practice- standard of care — All participating NICUs will be in the control arm during the first year prior to randomization to create a baseline of the current practices and between-units variation. NICUs in the control arm can continue conducting QI activities relevant to current practice, but without receiving the interventions outlined above until they transition to the intervention arm. The investigators will capture these activities and account for them in the analysis.
  Arms: Control Arm- Current management

SUMMARY:
The ABC-QI Trial aims to implement collaborative quality improvement (QI) strategies to standardize care for 32-36 week infants in Level 2 and 3 Neonatal intensive care units (NICUs) across the province of Alberta. The investigators want to know if using validated quality improvement methods and evidence-based care bundles will decrease the duration of hospital stay and get babies home as quickly as possible.

DETAILED DESCRIPTION:
A stepped-wedge cluster randomized trial will be conducted in 12 NICUs across Alberta (10 Level II and 2 Level III). Each NICU is considered a cluster and will be randomized to transition to the intervention arm at one of three time points.

The planned trial interventions include:

Intervention arm (Collaborative QI Strategies): The study intervention is a constellation of collaborative QI strategies: 1) QI Team Building; 2) QI Education; 3) Implementation of 2 standardized practice care bundles (Respiratory Care, and Nutritional Care); 4) QI mentoring; and 5) Collaborative networking. Based on the randomization, 4 NICUs will transition to the intervention arm at the end of each year.

Control arm (current management): All participating NICUs will be in the control arm during the first year prior to randomization to create a baseline of the current practices and between-units variation. NICUs in the control arm can continue conducting QI activities relevant to current practice, but without receiving the interventions outlined above.

ELIGIBILITY:
Inclusion Criteria:

Preterm Infants: Infants born at 32 to 36 weeks' gestation and admitted to the participating NICUs or postpartum units.

Quality Improvement Implementation Survey version 2 (QIIS-II) and semi-structured interview participants: Management staff, nurses, nurse practitioners, physicians, and allied health staff employed in participating NICUs.

Exclusion Criteria:

* Preterm Infants:

  * Major congenital anomalies or chromosomal abnormalities.
  * Primary admission to a surgical NICU: Alberta Children's Hospital or Stollery Children's Hospital.
  * Infants born in or transferred to a NICU outside Alberta.
  * Patients who have imposed confidentiality restrictions on accessing their health records.

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9500 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Length of Stay | Birth until discharge home or death, whichever came first, assessed until the participant reaches a corrected age of 6 months (6 months after their birth due date).
  The duration of hospitalization until final discharge.

SECONDARY OUTCOMES:
Cost to healthcare system per participant | Birth until discharge home or death, whichever came first, assessed until the participant reaches a corrected age of 6 months (6 months after their birth due date).
  The investigators will use the Canadian Institute for Health Information Patient Cost Estimator to calculate the daily cost based on the Case Mix Groups for gestational age and birth weight.
Number of participants with Hypothermia | Within 1 hour of birth
  Axillary temperature <36.5°C.
Number of participants with Hypoglycemia | First 24 hours of age
  Blood glucose <2.6 mmol/L.
Surfactant administration | First 168 hours of age.
  Date and method of administration
Duration of respiratory support | Birth until discharge home or death, whichever came first, assessed until the participant reaches a corrected age of 6 months (6 months after their birth due date).
  Total number of days administered
Age at achieving full enteral feeding | Birth until discharge home or death, whichever came first, assessed until the participant reaches a corrected age of 6 months (6 months after their birth due date).
  Date when the enteral intake reaches 120 ml/kg/day.
Time to regain birth weight | Birth until discharge home or death, whichever came first, assessed until the participant reaches a corrected age of 6 months (6 months after their birth due date).
  Difference in days between birth date and date when the infants regains or exceeds birth weight after initial weight loss.
Weight in grams | At discharge home in survivors, assessed up to a corrected age of 6 months (6 months after their birth due date).
  actual values in grams
Length in centimeters | At discharge home in survivors, assessed up to a corrected age of 6 months (6 months after their birth due date).
  actual values in centimeters
Head circumference in centimeters | At discharge home in survivors, assessed up to a corrected age of 6 months (6 months after their birth due date).
  actual values in centimeters
Breastmilk use | Birth until discharge home or death, whichever came first, assessed until the participant reaches a corrected age of 6 months (6 months after their birth due date).
  Defined as number of feeds where infant received breastfeeding or maternal expressed breastmilk
Number of unplanned rehospitalizations per participant | Within 30 days after discharge home
  Unplanned readmission to any hospital in Alberta following discharge
Number of emergency room visits per participant | Within 30 days after discharge home
  Emergency room visits to any hospital in Alberta following discharge
Hospital mortality | Until first discharge home, assessed until the participant reaches a corrected age of 6 months (6 months after their birth due date).
  Proportion of infants who dies before first discharge home
Infant mortality before 1 year of corrected age | Before 1 year of corrected age
  Corrected age = chronological age - days required for an infant to complete postmenstrual age of 40 weeks.
Transfer from Level II to Level III NICU | Until first discharge home, assessed until the participant reaches a corrected age of 6 months (6 months after their birth due date).
  Proportion of infants who require escalation of care and transfer to Level III NICU.
Staff perception of collaborative QI (EPIQ) implementation. | Year 2, 3, and 4 of study
  Semi-structured interviews with selected sample of staff from each NICU

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Abou Mehrem, MD, Principal Investigator — University of Calgary; Jennifer Toye, MD, Principal Investigator — University of Alberta
Locations (12):
- Canada (12):
  - Peter Lougheed Centre, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - Grande Prairie Regional Hospital, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Misericordia Community Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Sturgeon Community Hospital, Edmonton, Alberta
  - Chinook Regional Hospital, Lethbridge, Alberta
  - Medicine Hat Regional Hospital, Medicine Hat, Alberta
  - Red Deer Regional Hospital, Red Deer, Alberta

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, the de-identified, archived data will be transmitted to and stored at the Federated Research Data Repository (FRDR), for use by other researchers including those outside of the study.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after completion of the study and publication of the main manuscript.
Access Criteria: Approval from the principle investigator and the ABC-QI Trial Data Management Committee.

REFERENCES:
- [Derived] Abou Mehrem A, Toye J, Aziz K, Benzies K, Alshaikh B, Johnson D, Faris P, Soraisham A, McNeil D, Al Hamarneh YN, Foss K, Foulston C, Johns C, Zimmermann GL, Zein H, Hendson L, Kumaran K, Price D, Singhal N, Shah PS. Alberta Collaborative Quality Improvement Strategies to Improve Outcomes of Moderate and Late Preterm Infants (ABC-QI) Trial: a protocol for a multicentre, stepped-wedge cluster randomized trial. CMAJ Open. 2023 May 2;11(3):E397-E403. doi: 10.9778/cmajo.20220177. Print 2023 May-Jun. PMID 37130608